CLINICAL TRIAL: NCT01257542
Title: A Randomized, Parallel-Group, Double-Blind, Placebo-Controlled, Single-Dose, Pilot Study To Evaluate Efficacy Of Dextromethorphan Hydrobromide On Acute Cough In A Pediatric Population
Brief Title: Acute Cough Study In Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Collaborators: AccuDial Pharmaceutical, Inc. (Other); Boehringer Ingelheim (Industry); McNeil Consumer Healthcare Division of McNEIL-PPC, Inc. (Industry); Novartis (Industry); Perrigo Company (Industry); Procter and Gamble (Industry); Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6531001; RB-10-12
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Results first posted 2012-09-20 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-08

CONDITIONS: Common Cold; Infections, Upper Respiratory Tract
Keywords: randomized; parallel; double-blind; placebo-controlled; cough; efficacy; safety; dextromethorphan
MeSH Terms: conditions — Common Cold; Respiratory Tract Infections; Cough | interventions — Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: Dextromethorphan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan — A single 10 mL dose of Children's Triaminic Syrup (Dextromethorphan Hydrobromide 7.5 mg per 5 mL (total dose of 15 mg)
  Arms: Active
Drug: Placebo — A single 10 mL dose of matching placebo syrup
  Arms: Placebo

SUMMARY:
15 mg dextromethorphan hydrobromide will be better than placebo with respect to reducing the number of coughs over 6 hours and reducing the subjective severity of cough over 6 hours.

DETAILED DESCRIPTION:
In light of protocol changes required due to methodological and operational issues, including background noise in cough recordings which could impact data interpretation, the study has been terminated.

ELIGIBILITY:
Inclusion Criteria:

Male or female healthy children ages 6 to under 12 years who are symptomatic with a cough due to a cold or acute URTI characterized by:

* Onset of cold/URTI symptoms occurring no more than 10 days prior to Visit 1;
* At least 5 coughs during the second 30-minute period of the 60-minute baseline period.

General good health, aside from a common cold, and has no contraindications to the study or rescue medication

Exclusion Criteria:

* Acute, subchronic, or chronic cough due to any other condition other than a common cold

History of clinically significant cardiovascular, pulmonary, hepatic, renal, neurological, hematological, autoimmune, psychiatric, metabolic, gastro-intestinal or endocrine disease

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - DMI Research, Pinellas Park, Florida
  - Concentrics Center for Research, Indianapolis, Indiana
  - Cyn3rgy Research, Gresham, Oregon
  - Clinical Research Associates Incorporated, Nashville, Tennessee

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6531001&StudyName=Acute%20Cough%20Study%20In%20Children

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single oral dose of placebo solution matched to 15 milligram (mg) [10 milliliter (mL/)] dextromethorphan hydrobromide.
- Dextromethorphan Hydrobromide: Single oral dose of 15 mg (10 mL) dextromethorphan hydrobromide syrup [7.5 mg/5 milliliter (mL)].
Period: Overall Study
Arm/Group | Placebo | Dextromethorphan Hydrobromide
Started | 55 | 52
Completed | 52 | 45
Not Completed | 3 | 7
Not completed — Protocol Violation | 3 | 5
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dextromethorphan Hydrobromide | Total
Number analyzed (Participants) | 55 | 52 | 107
Age Continuous [Mean (Standard Deviation); unit: Years] | 8.9 (1.8) | 8.9 (1.6) | 8.9 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 25 | 57
  Male | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Total Cough Count
Description: Total cough count was done by trained assessors using continuous digital video and audio recordings.
Time Frame: Up to 6 hours post-dose
Population: Intent-to-treat (ITT) population included all randomized participants who received study medication, provided baseline efficacy data and any post baseline assessment.
Measure: Mean (Standard Deviation); unit: Cough counts
Arm/Group | Placebo | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 53 | 52
Cough counts | 238.7 (252.3) | 190.9 (190.6)
Statistical Analysis 1: Comparison: Placebo vs Dextromethorphan Hydrobromide; Odds Ratio and corresponding 95 percent (%) confidence interval (CI) were assessed from the negative binomial regression model; Test type: Superiority or Other; p = 0.252, Negative binomial regression — p-value was calculated using negative binomial regression model with treatment, site and baseline of cough count terms with log (exposure time) as the offset parameter; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.59 to 1.15]

2. Secondary Outcome: Change From Baseline in Perceived Verbal Cough Severity Scale for 6 Hour Post-Dose Period
Description: Perceived verbal cough severity score was assessed on a 5-point categorical rating scale in accordance to the question "How much have you coughed in the last hour?", where 0 = not at all, 1 = a tiny bit, 2 = a little, 3 = some and 4 = a lot. The change from baseline over the 6-hour post-dosing period calculated as the average of change from baseline [that is (i.e.) baseline value minus the post baseline value] measurements of Hour 1 to Hour 6, thus the change from baseline ranged from -4 to 4; higher score indicated a better improvement.
Time Frame: Baseline, 1, 2, 3, 4, 5, 6 hours post-dose
Population: ITT population included all randomized participants who received study medication, provided baseline efficacy data and any post baseline assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 53 | 52
Units on a scale
  Baseline | 3.0 (0.9) | 2.9 (0.9)
  Change for 6 hour post-dose period | 1.3 (1.1) | 1.1 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Dextromethorphan Hydrobromide; Treatment difference and corresponding 95% CI were calculated based on least-square (LS) means from analysis of variance (ANOVA) model; Test type: Superiority or Other; p = 0.134, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity verbal rating scale terms; LS mean difference = -0.26, 95% CI 2-sided [-0.60 to 0.08]

3. Secondary Outcome: Change From Baseline in Verbal Cough Severity Scale at Hours 1, 2, 3, 4, 5 and 6
Description: Verbal cough severity score was assessed on a 5-point categorical rating scale in accordance to the question "How much have you coughed in the last hour?", where 0 = not at all, 1 = a tiny bit, 2 = a little, 3 = some and 4 = a lot. The change from baseline values were derived by subtracting each post baseline value from the baseline value, and ranged from -4 to 4; higher score indicated a better improvement.
Time Frame: Baseline, 1, 2, 3, 4, 5, 6 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 53 | 52
Units on a scale
  Change at 1 hour | 1.0 (1.2) | 0.9 (1.2)
  Change at 2 hours | 1.2 (1.2) | 0.9 (1.4)
  Change at 3 hours | 1.3 (1.2) | 0.9 (1.4)
  Change at 4 hours | 1.4 (1.3) | 1.1 (1.4)
  Change at 5 hours | 1.7 (1.3) | 1.2 (1.4)
  Change at 6 hours | 1.5 (1.4) | 1.2 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Dextromethorphan Hydrobromide; 1 hour: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.768, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity verbal rating scale terms; LS mean difference = -0.06, 95% CI 2-sided [-0.45 to 0.33]
Statistical Analysis 2: Comparison: Placebo vs Dextromethorphan Hydrobromide; 2 hours: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.358, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity verbal rating scale terms; LS mean difference = -0.20, 95% CI 2-sided [-0.64 to 0.23]
Statistical Analysis 3: Comparison: Placebo vs Dextromethorphan Hydrobromide; 3 hours: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.139, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity verbal rating scale terms; LS mean difference = -0.32, 95% CI 2-sided [-0.74 to 0.10]
Statistical Analysis 4: Comparison: Placebo vs Dextromethorphan Hydrobromide; 4 hours: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.364, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity verbal rating scale terms; LS mean difference = -0.21, 95% CI 2-sided [-0.68 to 0.25]
Statistical Analysis 5: Comparison: Placebo vs Dextromethorphan Hydrobromide; 5 hours: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.039, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity verbal rating scale terms; LS mean difference = -0.46, 95% CI 2-sided [-0.90 to -0.02]
Statistical Analysis 6: Comparison: Placebo vs Dextromethorphan Hydrobromide; 6 hours: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.206, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity verbal rating scale terms; LS mean difference = -0.29, 95% CI 2-sided [-0.75 to 0.16]

4. Secondary Outcome: Change From Baseline in Perceived Numerical Cough Severity Scale for 6 Hour Post-Dose Period
Description: Perceived numerical cough severity score was assessed on an 11-point categorical rating scale in accordance to the question "How much have you coughed in the last hour?", where 0 = did not cough at all and 10 = cough a lot. The change from baseline for the 6-hour post-dosing period was calculated as the average of change from baseline (i.e. baseline value minus the post baseline value) measurements of Hour 1 to Hour 6, thus the change from baseline values ranged from -10 to 10; higher score indicated a better improvement.
Time Frame: Baseline, 1, 2, 3, 4, 5, 6 hour post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 53 | 52
Units on a scale
  Baseline | 6.8 (2.2) | 7.0 (2.3)
  Change for 6 hour post-dose period | 2.8 (2.5) | 2.5 (3.1)
Statistical Analysis 1: Comparison: Placebo vs Dextromethorphan Hydrobromide; Treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.304, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity numerical rating scale terms; LS mean difference = -0.49, 95% CI 2-sided [-1.43 to 0.45]

5. Secondary Outcome: Change From Baseline in Numerical Cough Severity Scale at Hours 1, 2, 3, 4, 5 and 6
Description: Numerical cough severity score was assessed on an 11-point categorical rating scale in accordance to the question "How much have you coughed in the last hour?", wherein 0 = did not cough at all and 10 = cough a lot. The change from baseline was derived by subtracting the post baseline value from the baseline value and ranged from -10 to 10; higher score indicated a better improvement.
Time Frame: Baseline, 1, 2, 3, 4, 5, 6 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 53 | 52
Units on a scale
  Change at 1 hour | 2.0 (2.9) | 2.0 (2.8)
  Change at 2 hours | 2.5 (2.6) | 2.1 (3.5)
  Change at 3 hours | 2.7 (2.7) | 2.3 (3.5)
  Change at 4 hours | 2.9 (2.8) | 2.5 (3.6)
  Change at 5 hours | 3.6 (2.8) | 3.0 (3.2)
  Change at 6 hours | 3.4 (3.3) | 2.8 (3.8)
Statistical Analysis 1: Comparison: Placebo vs Dextromethorphan Hydrobromide; 1 hour: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.954, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity numerical rating scale terms; LS mean difference = -0.03, 95% CI 2-sided [-1.03 to 0.97]
Statistical Analysis 2: Comparison: Placebo vs Dextromethorphan Hydrobromide; 2 hours: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.426, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity numerical rating scale terms; LS mean difference = -0.44, 95% CI 2-sided [-1.54 to 0.65]
Statistical Analysis 3: Comparison: Placebo vs Dextromethorphan Hydrobromide; 3 hours: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.396, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity numerical rating scale terms; LS mean difference = -0.45, 95% CI 2-sided [-1.49 to 0.60]
Statistical Analysis 4: Comparison: Placebo vs Dextromethorphan Hydrobromide; 4 hours: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.402, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity numerical rating scale terms; LS mean difference = -0.49, 95% CI 2-sided [-1.63 to 0.66]
Statistical Analysis 5: Comparison: Placebo vs Dextromethorphan Hydrobromide; 5 hours: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.204, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity numerical rating scale terms; LS mean difference = -0.69, 95% CI 2-sided [-1.75 to 0.38]
Statistical Analysis 6: Comparison: Placebo vs Dextromethorphan Hydrobromide; 6 hours: treatment difference and corresponding 95% CI were calculated based on LS means from ANOVA model; Test type: Superiority or Other; p = 0.179, ANOVA — p-value was calculated using ANOVA model with treatment, site and baseline cough severity numerical rating scale terms; LS mean difference = -0.84, 95% CI 2-sided [-2.06 to 0.39]

6. Secondary Outcome: Participants' Global Assessment of Cough: Cough Severity
Description: Participant global assessment of cough with the assistance of parent or legal guardian was scored on a 5-point categorical scale based on response to the question " How much have you coughed in the past 6 hours?" where 0 = not at all, 1 = a tiny bit, 2 = a little, 3 = some and 4 = a lot.
Time Frame: Within 5 minutes after Hour 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 53 | 52
Units on a scale | 3.1 (0.9) | 3.0 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Dextromethorphan Hydrobromide; Treatment difference and the associated 95% CI were based on the weighted Gamma statistics; Test type: Superiority or Other; p = 0.523, Cochran-Mantel-Haenszel — p-value was calculated from the Cochran-Mantel-Haenszel (CMH) test with modified ridit scores controlling site; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.21 to 0.39]

7. Secondary Outcome: Participants' Global Assessment of Cough: Relief From Cough
Description: Participant global assessment of cough with the assistance of parent or legal guardian was scored on a 5-point categorical scale based on response to the question "From when you woke up this morning until now, how much better is your cough?" where 0 = not at all better, 1 = a tiny bit better, 2 = a little better, 3 = better and 4 = a lot better.
Time Frame: Within 5 minutes after Hour 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Dextromethorphan Hydrobromide
Number analyzed (Participants) | 53 | 52
Units on a scale | 2.9 (1.0) | 2.7 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Dextromethorphan Hydrobromide; Treatment difference and the associated 95% CI were based on the weighted Gamma statistics; Test type: Superiority or Other; p = 0.796, Cochran-Mantel-Haenszel — p-value was calculated from the CMH test with modified ridit scores controlling site; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.35 to 0.24]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Dextromethorphan Hydrobromide
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/52
Other Adverse Events (participants affected / at risk) | 4/55 | 6/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=55) | Dextromethorphan Hydrobromide (N=52)
Nausea (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Headache (Nervous system disorders) | 0 | 3
Dizziness (Nervous system disorders) | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to methodological issues during study conduct, the study was terminated after only less than 50% of the targeted enrollment was achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.